CLINICAL TRIAL: NCT01582373
Title: Pilot Study to Assess the Efficacy of an Experimental 12-week Cognitive-behavioral Couple Therapy in the Treatment of Provoked Vestibulodynia
Brief Title: Pilot Study to Assess the Efficacy of Cognitive-behavioral Couple Therapy for Provoked Vestibulodynia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Sophie Bergeron, Associate professor, Université de Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBCT-01; 274271 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Vestibulodynia
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive-behavioral couple therapy (Experimental): The goals of CBCT are to enable participants to: (1) re-conceptualize PVD as a multidimensional pain problem influenced by a variety of factors including thoughts, emotions, behaviors and couple interactions; (2) re-conceptualize PVD as a couple problem in which both members of the couple affect and are affected by the pain; (3) modify those factors associated with pain during intercourse with a view to increasing adaptive coping, for example, by increasing self-efficacy and decreasing catastrophizing, as well as decreasing pain intensity; (4) improve the quality of their sexual functioning, reduce their sexual distress and increase their sexual satisfaction; (5) consolidate skills.
  Interventions: Behavioral: Cognitive-behavioral couple therapy

INTERVENTIONS:
Behavioral: Cognitive-behavioral couple therapy — The treatment package will include the following: information about the nature of CBCT; education about PVD and how it impacts on sexuality; education concerning a multifactorial view of pain; relaxation techniques; vaginal dilatation exercises; cognitive restructuring exercises (replacing distorted or irrational beliefs about pain and sexuality by more realistic ones); distraction techniques focusing on sexual imagery; expansion of the sexual repertoire; and exercises to improve pain and sexuality-relevant couple interactions (e.g., communication skills training, modification of maladaptive partner responses to pain, emotional disclosure and validation exercises).
  Other Names: Cognitive Behavioral Pain and Sex Therapy (CBPST)

SUMMARY:
The current pilot study aims to assess the feasibility and preliminary efficacy of a novel, 12-week targeted couple intervention (CBCT) for women with vulvodynia and their partners.

DETAILED DESCRIPTION:
Chronic pain problems involving the female reproductive system are major health concerns in women of all ages. As conditions which are poorly understood, they entail a great personal cost to patients and a significant financial cost to society. One such condition is vulvodynia, or chronic unexplained vulvar pain, which has a prevalence of 16%. Despite its negative impact on psychosexual and relationship satisfaction, there has been a paucity of research to provide empirically validated treatments for afflicted couples. The proposed research draws on findings from our work focusing on the influence of romantic relationships in the experience of vulvodynia as well as on our past studies evaluating the efficacy of group cognitive-behavioral therapy for this problem. The proposed pilot study aims to assess the feasibility and preliminary efficacy of a novel, 12-week targeted couple intervention (CBCT) for women with vulvodynia and their partners. The primary research question is: Is there a significant difference between pre- and post-treatment measures of pain during intercourse? We hypothesize that CBCT will yield pain reduction from pre- to post-treatment. The secondary research question focuses on pre- and post-treatment differences in 1) the multidimensional aspects of pain, 2) sexuality outcomes, 3) psychological adjustment, 4) relationship factors, and 5) patient self-reported improvement and treatment satisfaction. We hypothesize that the CBCT will result in significantly greater improvements on all outcome measures, and that the intervention will demonstrate adequate feasibility. Results of this study may improve the health and quality of life of patients afflicted with vulvodynia by helping us further develop this intervention for future clinical trial testing. For exploratory purposes, a 3-month follow-up assessment of treatment outcomes will also be conducted.

This pilot trial addresses the urgent need for empirically validated treatments for vulvodynia, and will help refine an intervention for future clinical trial testing. Results may improve the health and quality of life of couples afflicted with this highly prevalent women's health care problem. Findings will generate information about the feasibility and preliminary efficacy of a frequently recommended intervention for PVD, counselling targeting the couple. The findings will help provide women with PVD and their partners with scientifically based treatment options and may allow them to reduce the pain experienced during intercourse, in addition to improving their sexual functioning, overall well-being, and romantic relationship.

ELIGIBILITY:
Inclusion Criteria:

* pain during intercourse which is a) subjectively distressing, b) occurs on 80% of intercourse attempts, and c) has lasted for at least one year
* pain limited to intercourse and other activities involving pressure to the vestibule
* significant pain in one or more locations of the vestibule during the gynaecological exam, which is operationalized as a minimum average patient pain rating of 4 on a scale of 0 to 10
* having been sexually active as a couple in the last three months (intercourse, manual or oral stimulation)
* in a committed relationship for at least six months

Exclusion Criteria:

* vulvar pain not clearly linked to intercourse or pressure applied to the vestibule
* presence of one of the following: a) major medical and/or psychiatric illness, b) active infection, c) deep dyspareunia, d) vaginismus (as defined by DSM-IV), e) dermatologic lesion, f) pregnancy or planning a pregnancy
* age less than 18 or greater than 45

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pain during intercourse (Visual analog scale) | change in the VAS scores from pre- to post-treatment, and from pre-treatment to 3-month post-treatment
  Pain during intercourse will be assessed using a visual analog scale (VAS) ranging from 0 to 10, where 0 is no pain at all, and 10 is the worst pain ever. The main outcome will be the change in the VAS scores from pre- to post-treatment. This method for measuring pain has been shown to detect significant treatment effects in women with PVD and demonstrates a significant positive correlation with other pain intensity measures. Pain during intercourse is the main symptom of PVD and the one that most interferes with quality of life, hence the most relevant measure of functional outcome.

SECONDARY OUTCOMES:
Sexual function (Derogatis Interview for Sexual Functioning - Self-Report) | change in the DISF-SR scores from pre- to post-treatment, and from pre-treatment to 3-month post-treatment
  Sexual function will be assessed using the Derogatis Interview for Sexual Functioning - Self-Report (DISF-SR), which is a 25-item self-report version of a semi-structured interview designed to assess sexual function for both men and women. It measures five dimensions of sexuality: sexual cognition/fantasy, sexual arousal, sexual behavior/experience, orgasm, and sexual drive/relationship. Scores can be calculated for each dimension and for global sexual functioning. The DISF-SR boasts good internal consistency and reliability, specifically with women experiencing sexual dysfunction.
Global Measure of Sexual Satisfaction scale | change in GMSEX scores from pre-to post-treatment, and from pre-treatment to 3-month post-treatment
  Sexual satisfaction will be assessed using the Global Measure of Sexual Satisfaction scale, which consists of 5 items assessing global sexual satisfaction. Internal consistency of this scale is high (alpha = 0.90), as is test-retest reliability (r = 0.84) (Lawrance & Byers, 1998).
West Haven-Yale Multidimensional Pain Inventory - Significant Other Response Scale (MPI) | changes in MPI scores from pre- to post-treatment, and from pre-treatment to 3-month post-treatment
  Partner responses from the point of view of the women with PVD and their partners will be measured with the West Haven-Yale Multidimensional Pain Inventory - Significant Other Response Scale (MPI) (Kerns, Turk, & Rudy, 1985), and the Spouse Response Inventory - Facilitative subscale (SRI; (L. Schwartz, Mark P. Jensen, & Joan M. Romano, 2005) which have been adapted to our population of women with PVD and their partners.
Couple Satisfaction Index (CSI) | changes in CSI scores from pre- to post-treatment, and from pre-treatment to 3-month post-treatment
  Couple Satisfaction, or dyadic adjustment will be measured with the Couple Satisfaction Index (CSI). The CSI (Funk & Rogge, 2007) is a 32-item measure of relationship satisfaction. Compared to other well-known relationship satisfaction measures (e.g., Dyadic Adjustment Scale; Spanier, 1976; and the Marital Adjustment Test; Locke & Wallace, 1959) it demonstrates strong convergent validity, and a higher precision and power for detecting distinctions in satisfaction levels (Funk & Rogge, 2007).
Pain Catastrophizing Scale (PCS) | changes in PSC scores from pre-to post-treatment, and from pre-treatment to 3-month post-treatment
  Pain catastrophizing will be assessed using the Pain Catastrophizing Scale (Sullivan, Bishop, & Pivik, 1995), which consists of 13 items measuring exaggerated negative thoughts and feelings about the meaning of pain. Items are scored on a 5-point scale with the end points (0) not at all and (4) all the time. The PCS is a reliable and valid measure that has demonstrated a stable factorial structure across clinical and general populations, including a French population (French et al., 2005; Osman et al., 2000; Sullivan, et al., 1995).
Spielberger State-Trait Anxiety Inventory (STAI) | changes in STAI from pre-to post-treatment, and from pre-treatment to 3-month post-treatment
  Anxiety will be assessed using the Spielberger State-Trait Anxiety Inventory (STAI - (Spielberger, Gorsuch, & Lushene, 1970); ASTA - (Gauthier & Bouchard, 1993)). The STAI is a 40-item, well-known and widely used measure of state and trait anxiety that has demonstrated very good psychometric properties (Cronbach's alpha State = .93, Trait = .97) in various clinical and non-clinical samples including pain populations (Gauthier & Bouchard, 1993; Greenberg & Burns, 2003; Rule & Traver, 1983; Tanaka-Masumi & Kameoka, 1986).
Self-reported improvement and satisfaction | Reported at the end of treatment
  Patient self-reported improvement [scale of 0 (completely dissatisfied) to 10 (completely satisfied)] and treatment satisfaction [scale of 0 (worse) to 5 (complete cure)] will be measured at the post-treatment structured interview in order to assess the clinical significance of results.
Painful Intercourse Self-Efficacy Scale (PISES) | Changes in PISES scores from pre-to post-treatment, and from pre-treatment to 3-month post-treatment
  Pain self-efficacy will be assessed using the Painful Intercourse Self-Efficacy Scale (PISES; (Desrochers, et al., 2009), which was adapted from the Arthritis Self-Efficacy Scale (Lorig, Chastain, Ung, Shoor, & Holman, 1989). The PISES consists of 20 items with three subscales: self-efficacy for controlling pain during intercourse, self-efficacy for sexual function, and self-efficacy for controlling other symptoms.
Beck Depression Inventory (BDI-II) | changes in BDI-II scores from pre- to post-treatment, and from pre-treatment to 3-month post-treatment
  Depression or depression symptoms will be measured with the Beck Depression Inventory-II (BDI-II). The BDI-II is comprised of 21 items, with scores for most items ranging from 0 (low intensity) to 3 (high intensity) (Beck, Steer & Brown, 1996; Beck, Steer & Garvin, 1988). This measure of depression has been validated for use in chronic pain populations (Turner & Romano, 1984).

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Bergeron, PhD, Principal Investigator — Université de Montréal
Locations (1):
- Université de Montréal, Montreal, Quebec, Canada